CLINICAL TRIAL: NCT03742414
Title: SEAL (Stopping Eczema and ALlergy) Study: Prevent the Allergic March by Enhancing the Skin Barrier
Brief Title: Seal, Stopping Eczema and Allergy Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kari Nadeau, MD, PhD (Other)
Collaborators: National Jewish Health (Other); University of Chicago (Other); Children's Hospital Medical Center, Cincinnati (Other); Harvard School of Public Health (HSPH) (Other); Stanford University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); King's College London (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Kari Nadeau, MD, PhD, Chair, Department of Environmental Health, Harvard School of Public Health (HSPH)
Organization: Harvard School of Public Health (HSPH) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 48199; 1U01AI147462-01A1 (NIH)
Record Dates: First submitted 2018-10-30; First posted 2018-11-15 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-10

CONDITIONS: Eczema, Infantile; Eczema; Atopic Dermatitis Eczema; Atopic Dermatitis
Keywords: Dermatitis; Dry skin; Food allergy; Moisturizer
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Food Hypersensitivity | interventions — EpiCeram; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, parallel design trial designed for children (total n = 398) who have already developed atopic dermatitis (AD or eczema) by 12 weeks of age. The aim is to compare the effect of proactive sequential skin care, including the twice daily use of a tri-lipid skin barrier cream (Epiceram) or moisturizer and proactive use of fluticasone proprionate cream, against reactive AD therapy, to reduce the occurrence and severity of AD in early infancy and thereby prevent food allergy (FA).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Standard of care) (Active Comparator): The study doctors will provide standard of care with routine reactive topical products for atopic dermatitis flares
  Interventions: Other: Standard of Care
- Active Intervention arm (proactive treatment)- Epiceram (Experimental): Participants will receive proactive sequential skin care with the twice-daily use of a tri-lipid skin barrier cream (SBC). Clinically apparent eczema in this group will be managed with a short course of topical steroids (fluticasone propionate cream and/or hydrocortisone).
  Interventions: Combination Product: Tri-lipid skin barrier cream (Epiceram); Combination Product: Fluticasone propionate Cream 0.05%

INTERVENTIONS:
Combination Product: Tri-lipid skin barrier cream (Epiceram) — The aim is to compare the effect of proactive sequential skin care, including the twice daily use of a tri-lipid skin barrier cream (Epiceram) and proactive use of fluticasone proprionate cream, against reactive AD therapy, to reduce the occurrence and severity of AD in early infancy and thereby prevent food allergy (FA).
  Arms: Active Intervention arm (proactive treatment)- Epiceram
Combination Product: Fluticasone propionate Cream 0.05% — Proactive use of fluticasone proprionate cream for inflammation of the skin, to reduce the occurrence and severity of AD in early infancy and thereby prevent food allergy (FA).
  Arms: Active Intervention arm (proactive treatment)- Epiceram
Other: Standard of Care — Participants' eczema will be managed by their primary physician, i.e. standard of care with routine reactive topical products for atopic dermatitis flares.
  Arms: Control arm (Standard of care)

SUMMARY:
This is a randomized, controlled trial designed for children who are have already developed atopic dermatitis (AD or eczema) by 12 weeks of age. The aim is to compare the effect of proactive sequential skin care, including the twice-daily use of a tri-lipid skin barrier cream (Epiceram) and proactive use of fluticasone propionate cream, against reactive AD therapy, to reduce the occurrence and severity of AD in early infancy and thereby prevent food allergy (FA).

DETAILED DESCRIPTION:
This is a randomized, controlled, parallel design, open-label phase 2 clinical study to compare the efficacy of a proactive treatment arm versus the reactive arm, for the prevention of atopic dermatitis in children at high risk of food allergy. We will recruit 398 infants who have signs of dry skin or atopic dermatitis between 0-12 weeks of life.

The aim is to compare the effect of proactive sequential skin care, including the twice-daily use of a tri-lipid skin barrier cream (Epiceram) and proactive use of fluticasone propionate cream, against reactive AD therapy, to reduce the occurrence and severity of AD in early infancy and thereby prevent food allergy (FA).

ELIGIBILITY:
Inclusion Criteria:

1. Participants who develop early onset visible dry skin or atopic dermatitis up to and equal to 12 weeks of age.
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. In good general health as evidenced by medical history
4. No known adverse reaction to any of the study medications, their components or excipients

Exclusion Criteria:

1. Infants <3kg body weight
2. Infants with a chronic disease requiring therapy (e.g. heart disease, diabetes, serious neurological defects, immunodeficiency)
3. Known moderate to severe cutaneous skin disorder other than AD, including but not limited to cutaneous mastocytosis, bullous skin disease, pustular skin disease, neonatal HSV, aplasia, and albinism
4. Parents or guardians unwilling to sign consent
5. Current participant or participation since birth in any interventional study
6. Investigator or designee considers that the participant or parent/guardian would be unsuitable for inclusion in the study (for ex/ long stay in NICU)
7. A course of antibiotics in infant within 7 days of enrollment
8. Any known food allergies

Ages: 1 Week to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 398 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
number of foods each participant is sensitized to | 2 years
  Sensitization is defined as food-specific IgE > 0.1 kU/L

SECONDARY OUTCOMES:
The per-subject cumulative number of proven Food Allergy | 2 years
  Double-blind placebo-controlled oral food challenges used
Number of foods each participant is sensitized to | 24 months of age
  Sensitization is defined as food-specific skin prick test (SPT) ≥ 1 mm
Number of foods each participant is sensitized to | 24 months of age
  Sensitization is defined as food-specific skin prick test (SPT) ≥ 3 mm.
Presence, duration, and severity of dry skin and/or AD by clinical assessment | Baseline, 12, and 24 months of age and as necessary
  Patient-oriented SCORAD (PO-SCORAD) application used

CONTACTS AND LOCATIONS:
Overall Officials: Kari Nadeau, MD, PhD, Principal Investigator — Harvard
Locations (5):
- United States (4):
  - Sean N. Parker Center for Allergy & Asthma Research at Stanford University, Palo Alto, California
  - Division of Pediatric Allergy and Clinical Immunology, National Jewish Health, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
- • King's College London and Guy's and St. Thomas' NHS Foundation Trust, UK, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No current plan to share data

REFERENCES:
- See also: The Sean N. Parker Center for Allergy and Asthma Research at Stanford University — http://med.stanford.edu/allergyandasthma/about-us.html
- See also: SEAL study information — https://sealstudy.sites.stanford.edu/